CLINICAL TRIAL: NCT03797209
Title: A Post Market Survey to Detect Information of Adverse Events and Device Malfunctions of AXIOS Stent and Electrocautery Enhanced Delivery System Under Real World Medical Condition in Japan
Brief Title: Hot AXIOS System Japan Post Market Survey
Status: Completed | Type: Observational
Sponsor: Boston Scientific Japan K.K. (Industry)
Responsible Party: Sponsor
Other Study IDs: E7121
Record Dates: First submitted 2018-09-25; First posted 2019-01-09 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2022-03

CONDITIONS: Pancreatic Pseudocyst Infection; Pancreatic Pseudocyst; Walled Off Necrosis Infection; Walled Off Necrosis
Keywords: PPC; WON
MeSH Terms: conditions — Pancreatic Pseudocyst

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- AXIOS Patient
  Interventions: Device: EUS-guided fistulization AXIOS

INTERVENTIONS:
Device: EUS-guided fistulization AXIOS — By using a convex type ultrasonic endoscope to form a fistula by gastrointestinal puncture, to perform various drainage.

SUMMARY:
To detect information of Adverse Events and Device Malfunctions under real world medical condition in Japan.

ELIGIBILITY:
Inclusion Criteria:

* Patient who received implant procedure using study device at Japanese site.

Exclusion Criteria:

* NA

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient who received implant procedure using study device at Japanese site.
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
Safety (Adverse Events and Device Malfunction) | From implant procedure to 7 days after removal
Placement success | During implant procedure
  AXIOS stent is placed in an appropriate position using the delivery system.
Stent retention | From implant procedure to removal (a maximum of 60 days)
  AXIOS stent stays at the position where it was implanted during the implant procedure.
Stent lumen patency | From implant procedure to removal (a maximum of 60 days)
  The lumen of AXIOS stent is patent, and it can be used for drainage etc.
Decreased cyst size | From implant procedure to final observation (a maximum of 60 days)
Removal success | Removal procedure (a maximum of 60 days after implant procedure)
  AXIOS stent can be removed using standard endoscopic snares or forceps.

CONTACTS AND LOCATIONS:
Locations (40):
- Japan (40):
  - Aichi Medical University Hospital, Nagakute-Shi, Aichi-ken
  - Aichi Cancer Center Hospital, Nagoya, Aichi-ken
  - Nagoya University Hospital, Nagoya, Aichi-ken
  - Chiba University Hospital, Chiba, Chiba
  - Kameda Medical Center, Kamogawa-Shi, Chiba
  - National Cancer Center Hospital East, Kashiwa-Shi, Chiba
  - Tokyo Women's Medical University Yachiyo Medical Center, Yachiyo-Shi, Chiba
  - National Hospital Organization Kyushu Medical Center, Fukuoka, Fukuoka
  - Kyushu University Hospital, Fukuoka, Fukuoka
  - Teine Keijinkai Hospital, Sapporo, Hokkaido
  - Kobe University Hospital, Kobe, Hyōgo
  - Hyogo College of Medicine Hospital, Nishinomiya-Shi, Hyōgo
  - Kagoshima University Hospital, Kagoshima, Kagoshima-ken
  - Shonan Kamakura General Hospital, Kamakura-Shi, Kanagawa
  - Kitasato University Hospital, Sagamihara-Shi, Kanagawa
  - Yokohama Rosai Hospital, Yokohama, Kanagawa
  - Yokohama City University Medical Center, Yokohama, Kanagawa
  - Mie University Hospital, Tsu, Mie-ken
  - Tohoku University Hospital, Sendai, Miyagi
  - Sendai Open Hospital, Sendai, Miyagi
  - University of Miyazaki Hospital, Miyazaki, Miyazaki
  - Niigata University Medical and Dental Hospital, Niigata, Niigata
  - Kawasaki Medical School General Medical Center, Okayama, Okayama-ken
  - Okayama University Hospital, Okayama, Okayama-ken
  - Osaka City University Hospital, Osaka, Osaka
  - Kindai University Hospital, Osakasayama-Shi, Osaka
  - Osaka Medical College Hospital, Takatsuki-Shi, Osaka
  - Saitama Medical Universtity International Medical Center, Hidaka-Shi, Saitama
  - Saitama Medical Center, Kawagoe-Shi, Saitama
  - Kitasato University Medical Center, Kitamoto-Shi, Saitama
  - Tokyo Medical University Hospital, Tokyo, Shinjuku-Ku
  - Jichi Medical University Hospital, Shimotsuke-Shi, Tochigi
  - Saiseikai Utsunomiya Hospital, Utsunomiya, Tochigi
  - Juntendo University Hospital, Bunkyo-Ku, Tokyo
  - Toho University Ohashi Medical Center, Meguro-Ku, Tokyo
  - The Jikei University Hospital, Minato-Ku, Tokyo
  - Kyorin University Hospital, Mitaka-Shi, Tokyo
  - Keio University Hospital, Shinjuku-Ku, Tokyo
  - Tokyo Women's Medical University Hospital, Shinjuku-Ku, Tokyo
  - Wakayama Medical University Hospital, Wakayama, Wakayama

IPD SHARING:
Plan to Share IPD: No